CLINICAL TRIAL: NCT00097786
Title: A Multinational, Randomized, Double-blind, Placebo-controlled, Forced-titration, 2 x 2 Factorial Design Study of the Efficacy and Safety of Long-term Administration of Nateglinide and Valsartan in the Prevention of Diabetes and Cardiovascular Outcomes in Subjects With Impaired Glucose Tolerance (IGT)
Brief Title: Long-term Study of Nateglinide+Valsartan to Prevent or Delay Type II Diabetes Mellitus and Cardiovascular Complications
Acronym: Navigator
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Study Director, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: CDJN608B2302
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Prevention; Diabetes type 2; valsartan; nateglinide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Valsartan; Nateglinide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Valsartan 160 mg + nateglinide 60 mg (Experimental): For the first 2 weeks of treatment, patients took the combination of nateglinide 30 mg (3 times daily, ante cibum [ac] before meals) and valsartan 80 mg (once daily [od] in the morning). After 2 weeks, patients were up-titrated to nateglinide 60 mg ac and valsartan 160 mg od.
  Interventions: Drug: Valsartan 160 mg + nateglinide 60 mg
- Valsartan 160 mg + nateglinide placebo (Experimental): For the first 2 weeks of treatment, patients took valsartan 80 mg capsules (once daily [od] in the morning). After 2 weeks, patients were up-titrated to 160 mg valsartan od. Patients also received nateglinide placebo tablets (3 times daily, ante cibum [ac] before meals).
  Interventions: Drug: Valsartan 160 mg + nateglinide placebo
- Nateglinide 60 mg + valsartan placebo (Experimental): For the first 2 weeks of treatment, patients took nateglinide 30 mg tablets (3 times daily, ante cibum [ac] before meals). After 2 weeks, patients were uptitrated to 60 mg nateglinide ac. Patients also received valsartan placebo capsules (once daily [od] in the morning).
  Interventions: Drug: Nateglinide 60 mg + valsartan placebo
- Placebo (Placebo Comparator): Patients took 3 nateglinide placebo tablets (3 times daily, ante cibum [ac] before meals) and 1 valsartan placebo capsule (once daily [od] in the morning).
  Interventions: Drug: Valsartan placebo + nateglinide placebo

INTERVENTIONS:
Drug: Valsartan 160 mg + nateglinide 60 mg — The double-blinding of the randomized study medication was maintained by the use of identical placebo and active tablets and capsules for nateglinide and valsartan, respectively. Patients were instructed not to take the morning dose of either medication nor to eat breakfast on the day of a scheduled study visit, but to wait until after the visit was completed. Patients not tolerating the higher dose (Level 2) were down-titrated to receive Level 1. Patients not tolerating the lower dose (Level 1) had a treatment interruption. Starting at Week 2 and throughout the study, attempts were to be made to reach the highest dose level (Level 2), if medically acceptable. Following each change in dose level or re-initiation of treatment, tolerability was assessed after 2 weeks of exposure.
  Arms: Valsartan 160 mg + nateglinide 60 mg
Drug: Valsartan 160 mg + nateglinide placebo — The double-blinding of the randomized study medication was maintained by the use of identical placebo and active tablets and capsules for nateglinide and valsartan, respectively. Patients were instructed not to take the morning dose of either medication nor to eat breakfast on the day of a scheduled study visit, but to wait until after the visit was completed. Patients not tolerating the higher dose (Level 2) were down-titrated to receive Level 1. Patients not tolerating the lower dose (Level 1) had a treatment interruption. Starting at Week 2 and throughout the study, attempts were to be made to reach the highest dose level (Level 2), if medically acceptable. Following each change in dose level or re-initiation of treatment, tolerability was assessed after 2 weeks of exposure.
  Arms: Valsartan 160 mg + nateglinide placebo
Drug: Nateglinide 60 mg + valsartan placebo — The double-blinding of the randomized study medication was maintained by the use of identical placebo and active tablets and capsules for nateglinide and valsartan, respectively. Patients were instructed not to take the morning dose of either medication nor to eat breakfast on the day of a scheduled study visit, but to wait until after the visit was completed. Patients not tolerating the higher dose (Level 2) were down-titrated to receive Level 1. Patients not tolerating the lower dose (Level 1) had a treatment interruption. Starting at Week 2 and throughout the study, attempts were to be made to reach the highest dose level (Level 2), if medically acceptable. Following each change in dose level or re-initiation of treatment, tolerability was assessed after 2 weeks of exposure.
  Arms: Nateglinide 60 mg + valsartan placebo
Drug: Valsartan placebo + nateglinide placebo — The double-blinding of the randomized study medication was maintained by the use of identical placebo and active tablets and capsules for nateglinide and valsartan, respectively. Patients were instructed not to take the morning dose of either medication nor to eat breakfast on the day of a scheduled study visit, but to wait until after the visit was completed. Patients not tolerating the higher dose (Level 2) were down-titrated to receive Level 1. Patients not tolerating the lower dose (Level 1) had a treatment interruption. Starting at Week 2 and throughout the study, attempts were to be made to reach the highest dose level (Level 2), if medically acceptable. Following each change in dose level or re-initiation of treatment, tolerability was assessed after 2 weeks of exposure.
  Arms: Placebo

SUMMARY:
This study is a test of the safety and effectiveness of two drugs, one for diabetes and one for hypertension, in keeping patients with high lab values of glucose from progressing to frank diabetes and developing cardiovascular complications. People in this study cannot have frank diabetes but are considered "borderline" based on blood tests. People in the study take none, one or both of the drugs and do not know which one(s) they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Impaired glucose tolerance
* Age dependent risk factors

Exclusion Criteria:

* Frank diabetes

For detailed information, call contact person.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9306 (Actual)
Dates: Start 2002-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- Multiple Locations, New Jersey, United States
- Investigative Site, Argentina
- Investigative Site, Australia
- Multiple Locations, Austria
- Investigative Site, Belgium
- Investigative Site, Brazil
- Investigative Site, Canada
- Investigative Site, Chile
- Investigative Site, China
- Investigative Site, Colombia
- Investigative Site, Czechia
- Investigative Site, Denmark
- Investigative Site, Ecuador
- Investigative Site, Finland
- Investigative Site, France
- Investigative Site, Germany
- Investigative Site, Greece
- Investigative Site, Guatemala
- Investigative Site, Hong Kong
- Investigative Site, Hungary
- Investigative Site, Italy
- Investigative Site, Malaysia
- Investigative Site, Mexico
- Investigative Site, Netherlands
- Investigative Site, Norway
- Investigative Site, Peru
- Investigative Site, Poland
- Investigative Site, Russia
- Investigative Site, Singapore
- Investigative Site, Slovakia
- Investigative Site, South Africa
- Investigative Site, Spain
- Investigative Site, Sweden
- Investigative Site, Switzerland
- Investigative Site, Taiwan
- Investigative Site, Turkey (Türkiye)
- Investigative Site, United Kingdom
- Investigative Site, Uruguay

REFERENCES:
- [Derived] Harumi Higuchi Dos Santos M, Sharma A, Sun JL, Pieper K, McMurray JJ, Holman RR, Lopes RD. International Variation in Outcomes Among People with Cardiovascular Disease or Cardiovascular Risk Factors and Impaired Glucose Tolerance: Insights from the NAVIGATOR Trial. J Am Heart Assoc. 2017 Jan 13;6(1):e003892. doi: 10.1161/JAHA.116.003892. PMID 28087508
- [Derived] Preiss D, Thomas LE, Wojdyla DM, Haffner SM, Gill JM, Yates T, Davies MJ, Holman RR, McMurray JJ, Califf RM, Kraus WE; NAVIGATOR Investigators. Prospective relationships between body weight and physical activity: an observational analysis from the NAVIGATOR study. BMJ Open. 2015 Aug 14;5(8):e007901. doi: 10.1136/bmjopen-2015-007901. PMID 26275900
- [Derived] Katz M, Califf RM, Sun JL, McMurray JJ, Thomas L, Lopes RD. Venous thromboembolism and cardiovascular risk: results from the NAVIGATOR trial. Am J Med. 2015 Mar;128(3):297-302. doi: 10.1016/j.amjmed.2014.08.022. Epub 2014 Nov 20. PMID 25447626
- [Derived] Preiss D, Haffner SM, Thomas LE, Sun JL, Sattar N, Yates T, J Davies M, McMurray JJ, Holman RR, Califf RM, Kraus WE. Change in levels of physical activity after diagnosis of type 2 diabetes: an observational analysis from the NAVIGATOR study. Diabetes Obes Metab. 2014 Dec;16(12):1265-8. doi: 10.1111/dom.12320. Epub 2014 Jun 19. PMID 24861892
- [Derived] Huffman KM, Sun JL, Thomas L, Bales CW, Califf RM, Yates T, Davies MJ, Holman RR, McMurray JJ, Bethel MA, Tuomilehto J, Haffner SM, Kraus WE. Impact of baseline physical activity and diet behavior on metabolic syndrome in a pharmaceutical trial: results from NAVIGATOR. Metabolism. 2014 Apr;63(4):554-61. doi: 10.1016/j.metabol.2014.01.002. Epub 2014 Jan 15. PMID 24559843
- [Derived] Yates T, Haffner SM, Schulte PJ, Thomas L, Huffman KM, Bales CW, Califf RM, Holman RR, McMurray JJ, Bethel MA, Tuomilehto J, Davies MJ, Kraus WE. Association between change in daily ambulatory activity and cardiovascular events in people with impaired glucose tolerance (NAVIGATOR trial): a cohort analysis. Lancet. 2014 Mar 22;383(9922):1059-66. doi: 10.1016/S0140-6736(13)62061-9. Epub 2013 Dec 20. PMID 24361242
- [Derived] Shen L, Shah BR, Reyes EM, Thomas L, Wojdyla D, Diem P, Leiter LA, Charbonnel B, Mareev V, Horton ES, Haffner SM, Soska V, Holman R, Bethel MA, Schaper F, Sun JL, McMurray JJ, Califf RM, Krum H. Role of diuretics, beta blockers, and statins in increasing the risk of diabetes in patients with impaired glucose tolerance: reanalysis of data from the NAVIGATOR study. BMJ. 2013 Dec 9;347:f6745. doi: 10.1136/bmj.f6745. PMID 24322398
- [Derived] NAVIGATOR Study Group; McMurray JJ, Holman RR, Haffner SM, Bethel MA, Holzhauer B, Hua TA, Belenkov Y, Boolell M, Buse JB, Buckley BM, Chacra AR, Chiang FT, Charbonnel B, Chow CC, Davies MJ, Deedwania P, Diem P, Einhorn D, Fonseca V, Fulcher GR, Gaciong Z, Gaztambide S, Giles T, Horton E, Ilkova H, Jenssen T, Kahn SE, Krum H, Laakso M, Leiter LA, Levitt NS, Mareev V, Martinez F, Masson C, Mazzone T, Meaney E, Nesto R, Pan C, Prager R, Raptis SA, Rutten GE, Sandstroem H, Schaper F, Scheen A, Schmitz O, Sinay I, Soska V, Stender S, Tamas G, Tognoni G, Tuomilehto J, Villamil AS, Vozar J, Califf RM. Effect of valsartan on the incidence of diabetes and cardiovascular events. N Engl J Med. 2010 Apr 22;362(16):1477-90. doi: 10.1056/NEJMoa1001121. Epub 2010 Mar 14. PMID 20228403
- [Derived] NAVIGATOR Study Group; Holman RR, Haffner SM, McMurray JJ, Bethel MA, Holzhauer B, Hua TA, Belenkov Y, Boolell M, Buse JB, Buckley BM, Chacra AR, Chiang FT, Charbonnel B, Chow CC, Davies MJ, Deedwania P, Diem P, Einhorn D, Fonseca V, Fulcher GR, Gaciong Z, Gaztambide S, Giles T, Horton E, Ilkova H, Jenssen T, Kahn SE, Krum H, Laakso M, Leiter LA, Levitt NS, Mareev V, Martinez F, Masson C, Mazzone T, Meaney E, Nesto R, Pan C, Prager R, Raptis SA, Rutten GE, Sandstroem H, Schaper F, Scheen A, Schmitz O, Sinay I, Soska V, Stender S, Tamas G, Tognoni G, Tuomilehto J, Villamil AS, Vozar J, Califf RM. Effect of nateglinide on the incidence of diabetes and cardiovascular events. N Engl J Med. 2010 Apr 22;362(16):1463-76. doi: 10.1056/NEJMoa1001122. Epub 2010 Mar 14. PMID 20228402
- [Derived] Krum H, McMurray JJ, Horton E, Gerlock T, Holzhauer B, Zuurman L, Haffner SM, Bethel MA, Holman RR, Califf RM. Baseline characteristics of the Nateglinide and Valsartan Impaired Glucose Tolerance Outcomes Research (NAVIGATOR) trial population: comparison with other diabetes prevention trials. Cardiovasc Ther. 2010 Apr;28(2):124-32. doi: 10.1111/j.1755-5922.2010.00146.x. Epub 2010 Feb 23. PMID 20184589
- [Derived] Bethel MA, Deedwania P, Levitt NS, Schmitz O, Huntsman-Labed A, Califf RM, Haffner SM, Diem P; NAVIGATOR Study Group. Metabolic syndrome and alanine aminotransferase: a global perspective from the NAVIGATOR screening population. Diabet Med. 2009 Dec;26(12):1204-11. doi: 10.1111/j.1464-5491.2009.02864.x. PMID 20002471
- [Derived] Bethel MA, Holman R, Haffner SM, Califf RM, Huntsman-Labed A, Hua TA, McMurray J. Determining the most appropriate components for a composite clinical trial outcome. Am Heart J. 2008 Oct;156(4):633-40. doi: 10.1016/j.ahj.2008.05.018. Epub 2008 Jul 31. PMID 18926145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially enrolled 9518, 212 excluded.
Groups:
- Valsartan 160 mg od + Nateglinide 60 mg ac: For the first 2 weeks of treatment, patients took the combination of nateglinide 30 mg (3 times daily ante cibum [ac, before meals]) and valsartan 80 mg (once daily [od] in the morning). After 2 weeks, patients were uptitrated to nateglinide 60 mg ac and valsartan 160 mg od.
- Valsartan 160 mg od + Placebo Nateglinide: For the first 2 weeks of treatment, patients took valsartan 80 mg once daily (od) once in the morning. After 2 weeks, patients were uptitrated to 160 mg valsartan od. Patient also received placebo matching nateglinide tablets identical to the active nateglinide tablets (ac, before meals).
- Nateglinide 60 mg ac + Placebo Valsartan: For the first 2 weeks of treatment, patients took one 30 mg tablet of nateglinide with a glass of water 1-30 minutes before each main meal of the day, ie, 3 times daily ante cibum (ac, before meals). If a meal was missed, the patient was not to take a tablet. After 2 weeks, patients were uptitrated to 60 mg nateglinide ac. Patients also received placebo matching valsartan capsules identical to the active valsartan capsules.
- Placebo: Patients took 3 placebo tablets identical to nateglinide tablets 3 times daily ac and 1 placebo capsule identical to valsartan capsule once daily in the morning.
Period: Overall Study
Arm/Group | Valsartan 160 mg od + Nateglinide 60 mg ac | Valsartan 160 mg od + Placebo Nateglinide | Nateglinide 60 mg ac + Placebo Valsartan | Placebo
Started | 2316 ("Started" indicates Full Analysis Set (FAS) population. Initially enrolled 9518, 212 excluded.) | 2315 | 2329 | 2346
Complete FU for Progression to Diabetes | 1709 | 1712 | 1734 | 1762
Complete Follow-up for Extended CV EPs | 1969 | 1985 | 1987 | 2015
Complete Follow-up for Core CV EPs | 1948 | 1963 | 1966 | 1988
Completed | 2020 ("Completed" means completed follow up for all cause death.) | 2023 | 2016 | 2036
Not Completed | 296 | 292 | 313 | 310
Not completed — lost to follow-up for all-cause death | 296 | 292 | 313 | 310

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan 160 mg od + Nateglinide 60 mg ac | Valsartan 160 mg od + Placebo Nateglinide | Nateglinide 60 mg ac + Placebo Valsartan | Placebo | Total
Number analyzed (Participants) | 2316 | 2315 | 2329 | 2346 | 9306
Age, Continuous [Mean (Standard Deviation); unit: years] — Originally 9518 patient were enrolled and 212 excluded. So this baseline measure is based on Full analysis Set(FAS)population.
  years | 63.7 (6.75) | 63.7 (6.91) | 63.8 (6.82) | 63.9 (6.88) | 63.8 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants] — Originally 9518 patient were enrolled and 212 excluded. So this baseline measure is based on Full analysis Set(FAS)population.
  Participants
    Female | 1174 | 1140 | 1194 | 1203 | 4711
    Male | 1142 | 1175 | 1135 | 1143 | 4595

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Reaching the Endpoint: Progression to Diabetes - Valsartan Versus Non-valsartan
Description: Progression to diabetes was determined by (a) an algorithm based on central laboratory measurements of fasting plasma glucose and/or a 2 hour oral glucose tolerance test or (b) adjudication by the Diabetes Endpoint Adjudication Committee.
Time Frame: Mean patient duration of 4.2 years
Population: Full Analysis Set: All patients in the randomized set with the exception of patients from 10 Mexican sites closed for severe Good Clinical Practice deficiencies.
Measure: Number; unit: Percentage of patients
Groups:
- Valsartan: All patients from the treatment arms (1) combined valsartan 160 mg od and nateglinide 60 mg ac and (2) valsartan 160 mg od only.
- Non-valsartan: All patients from the treatment arms (1) nateglinide 60 mg ac and (2) placebo.
Arm/Group | Valsartan | Non-valsartan
Number analyzed (Participants) | 4631 | 4675
Percentage of patients | 33.1 | 36.8

2. Primary Outcome: Percentage of Patients Reaching the Endpoint: Extended Morbidity and Mortality Event - Valsartan Versus Non-valsartan
Description: The extended cardiovascular endpoint was defined as a cardiovascular morbidity/mortality event including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, revascularization procedure, hospitalization for congestive heart failure, and hospitalization for unstable angina.
Time Frame: Mean patient duration of 5.6 years
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan | Non-valsartan
Number analyzed (Participants) | 4631 | 4675
Percentage of patients | 14.5 | 14.8

3. Primary Outcome: Percentage of Patients Reaching the Endpoint: Core Cardiovascular Morbidity and Mortality Event - Valsartan Versus Non-valsartan
Description: The core cardiovascular endpoint was defined as a cardiovascular morbidity/mortality event including cardiovascular death, non-fatal myocardial infarction, non-fatal stroke and hospitalization for congestive heart failure.
Time Frame: Mean patient duration of 5.8 years
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan | Non-valsartan
Number analyzed (Participants) | 4631 | 4675
Percentage of patients | 8.1 | 8.1

4. Primary Outcome: Percentage of Patients Reaching the Endpoint: Progression to Diabetes - Nateglinide Versus Non-nateglinide
Description: as for outcome 1
Time Frame: Mean patient duration of 4.2 years
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Groups:
- Nateglinide: All patients from the treatment arm (1) combined valsartan 160 mg od and nateglinide 60 mg ac and (2) nateglinide 60 mg ac only.
- Non-nateglinide: All patients from the treatment arms (1) valsartan 160 mg od and (2) placebo.
Arm/Group | Nateglinide | Non-nateglinide
Number analyzed (Participants) | 4645 | 4661
Percentage of patients | 36.0 | 33.9

5. Primary Outcome: Percentage of Patients Reaching the Endpoint: Extended Morbidity and Mortality Event - Nateglinide Versus Non-nateglinide
Description: as for outcome 2
Time Frame: Mean patient duration of 5.6 years
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Nateglinide | Non-nateglinide
Number analyzed (Participants) | 4645 | 4661
Percentage of patients | 14.2 | 15.2

6. Primary Outcome: Percentage of Patients Reaching the Endpoint: Core Cardiovascular Morbidity and Mortality Event - Nateglinide Versus Non-nateglinide
Description: as for outcome 3
Time Frame: Mean patient duration of 5.8 years
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Nateglinide | Non-nateglinide
Number analyzed (Participants) | 4645 | 4661
Percentage of patients | 7.9 | 8.3

ADVERSE EVENTS:
Time Frame: The maximum follow-up time was 7.7 years with the mean follow-up time of approximately 6 years.
Description: Patients were recruited over a two year period and were followed for Adverse Event reporting until the target number of patients had experienced an extended cardiovascular endpoint. Hence, the follow-up time was not the same for all patients.
Arm/Group | Valsartan 160 mg od + Nateglinide 60 mg ac | Valsartan 160 mg od + Placebo Nateglinide | Nateglinide 60 mg ac + Placebo Valsartan | Placebo
Serious Adverse Events (participants affected / at risk) | 1031/2297 | 1040/2283 | 1035/2305 | 1049/2316
Other Adverse Events (participants affected / at risk) | 1970/2297 | 1932/2283 | 1951/2305 | 1934/2316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 160 mg od + Nateglinide 60 mg ac (N=2297) | Valsartan 160 mg od + Placebo Nateglinide (N=2283) | Nateglinide 60 mg ac + Placebo Valsartan (N=2305) | Placebo (N=2316)
Anaemia (Blood and lymphatic system disorders) | 19 | 10 | 18 | 19
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 2
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Accelerated idioventricular rhythm (Cardiac disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 12 | 8 | 13 | 9
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 27 | 32 | 23 | 21
Angina pectoris (Cardiac disorders) | 92 | 99 | 71 | 74
Angina unstable (Cardiac disorders) | 46 | 63 | 61 | 60
Aortic valve disease (Cardiac disorders) | 1 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 4 | 1 | 3 | 3
Aortic valve stenosis (Cardiac disorders) | 1 | 2 | 3 | 1
Arrhythmia (Cardiac disorders) | 13 | 12 | 8 | 8
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 1 | 2 | 3
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 60 | 46 | 57 | 63
Atrial flutter (Cardiac disorders) | 8 | 3 | 7 | 5
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 3
Atrioventricular block complete (Cardiac disorders) | 3 | 7 | 5 | 2
Atrioventricular block first degree (Cardiac disorders) | 1 | 1 | 0 | 3
Atrioventricular block second degree (Cardiac disorders) | 2 | 2 | 5 | 1
Atrioventricular dissociation (Cardiac disorders) | 0 | 0 | 0 | 1
Bifascicular block (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 9 | 10 | 11 | 9
Bundle branch block (Cardiac disorders) | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 3 | 1 | 2 | 1
Bundle branch block right (Cardiac disorders) | 0 | 3 | 1 | 0
Cardiac arrest (Cardiac disorders) | 11 | 6 | 8 | 3
Cardiac asthma (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 16 | 26 | 16 | 18
Cardiac failure acute (Cardiac disorders) | 1 | 3 | 2 | 3
Cardiac failure chronic (Cardiac disorders) | 2 | 4 | 3 | 3
Cardiac failure congestive (Cardiac disorders) | 22 | 32 | 37 | 35
Cardiac fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 4 | 5 | 1
Cardiogenic shock (Cardiac disorders) | 2 | 2 | 5 | 2
Cardiomegaly (Cardiac disorders) | 1 | 0 | 2 | 2
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 2 | 3 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 2 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 3 | 1 | 1 | 2
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 43 | 37 | 50 | 42
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 2 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 8 | 10 | 6 | 9
Coronary artery perforation (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 15 | 10 | 7 | 12
Coronary artery thrombosis (Cardiac disorders) | 2 | 0 | 1 | 0
Coronary ostial stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Dilatation ventricular (Cardiac disorders) | 1 | 0 | 0 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 2 | 1 | 0
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 3 | 3 | 1
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 3 | 4 | 0
Left ventricular failure (Cardiac disorders) | 4 | 3 | 4 | 6
Left ventricular hypertrophy (Cardiac disorders) | 3 | 0 | 1 | 1
Microvascular angina (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 4 | 2 | 4
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 1 | 1 | 1
Myocardial infarction (Cardiac disorders) | 46 | 41 | 46 | 46
Myocardial ischaemia (Cardiac disorders) | 20 | 17 | 22 | 19
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 6 | 3 | 4 | 7
Pericardial effusion (Cardiac disorders) | 4 | 2 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1 | 3
Postinfarction angina (Cardiac disorders) | 1 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0 | 1
Reperfusion arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 6 | 4 | 11 | 11
Silent myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 2 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 2 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 8 | 3 | 8 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 4 | 0 | 3
Subendocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 2 | 2
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 4 | 3 | 5 | 5
Tachyarrhythmia (Cardiac disorders) | 0 | 3 | 0 | 0
Tachycardia (Cardiac disorders) | 4 | 6 | 5 | 6
Tricuspid valve incompetence (Cardiac disorders) | 2 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 6 | 5 | 3
Ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 6 | 6 | 2 | 2
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 5 | 12 | 6
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Myocardial bridging (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear canal stenosis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 5 | 6 | 4
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 3
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 3 | 1
Adrenal cyst (Endocrine disorders) | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 1
Adrenal mass (Endocrine disorders) | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 2 | 1 | 0 | 0
Goitre (Endocrine disorders) | 7 | 8 | 2 | 2
Hyperparathyroidism (Endocrine disorders) | 1 | 1 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 2 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 5 | 4 | 2 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 | 0 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 1 | 1 | 0 | 0
Secondary hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 1
Thyroid disorder (Endocrine disorders) | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 2 | 1 | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Blindness transient (Eye disorders) | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 2
Cataract (Eye disorders) | 9 | 19 | 10 | 17
Cataract nuclear (Eye disorders) | 0 | 1 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 2 | 1
Endocrine ophthalmopathy (Eye disorders) | 0 | 0 | 0 | 1
Exophthalmos (Eye disorders) | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 3 | 1 | 3 | 0
Hyalosis asteroid (Eye disorders) | 0 | 0 | 0 | 1
Lens dislocation (Eye disorders) | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 1
Macular hole (Eye disorders) | 1 | 1 | 0 | 0
Maculopathy (Eye disorders) | 0 | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 0 | 1 | 0 | 0
Panophthalmitis (Eye disorders) | 0 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 2
Retinal detachment (Eye disorders) | 0 | 3 | 6 | 3
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal ischaemia (Eye disorders) | 0 | 1 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 1 | 0
Retinal vascular thrombosis (Eye disorders) | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 0 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 4 | 5 | 4 | 4
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 18 | 13 | 15 | 15
Abdominal pain lower (Gastrointestinal disorders) | 0 | 4 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 15 | 5 | 4 | 4
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal polyp (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal prolapse (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 5 | 1 | 2
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bezoar (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 5 | 7 | 1 | 5
Constipation (Gastrointestinal disorders) | 6 | 3 | 1 | 4
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 7 | 9 | 11
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 6 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 5 | 3 | 3 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Duodenal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2 | 4 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1 | 2 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Enterocele (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Enterocolonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 4 | 0 | 5
Gastric polyps (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 5 | 4 | 2 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2 | 3 | 4
Gastric volvulus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 8 | 6 | 8 | 6
Gastritis erosive (Gastrointestinal disorders) | 4 | 1 | 2 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 9 | 12 | 11
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Gastrolithiasis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 6 | 4 | 2
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 4 | 5 | 6
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 3 | 4 | 2 | 6
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 5 | 2 | 1 | 5
Ileus paralytic (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 18 | 22 | 22 | 22
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 4 | 4 | 5
Intestinal perforation (Gastrointestinal disorders) | 3 | 1 | 2 | 2
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Intestinal strangulation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Ischiorectal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Large intestinal stricture (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 4 | 1 | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 10 | 9 | 9
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 9 | 2 | 3 | 6
Pancreatitis acute (Gastrointestinal disorders) | 7 | 3 | 6 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Papilla of Vater stenosis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 5 | 4 | 3 | 3
Polyp colorectal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 5 | 6 | 8
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 1 | 1 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1 | 3 | 1
Subileus (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 4 | 7 | 4 | 4
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3 | 2 | 4
Vomiting (Gastrointestinal disorders) | 14 | 15 | 10 | 9
Asthenia (General disorders) | 4 | 6 | 6 | 8
Cardiac death (General disorders) | 1 | 0 | 0 | 0
Catheter related complication (General disorders) | 0 | 1 | 1 | 0
Catheter thrombosis (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 3 | 2 | 3 | 3
Chest pain (General disorders) | 15 | 6 | 10 | 12
Chills (General disorders) | 0 | 2 | 1 | 1
Chronic fatigue syndrome (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 10 | 19 | 11 | 14
Exercise tolerance decreased (General disorders) | 1 | 0 | 1 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0
Fat necrosis (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 1
Foreign body reaction (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 1 | 4 | 0
General physical health deterioration (General disorders) | 3 | 1 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 2 | 1 | 0
Hernia obstructive (General disorders) | 1 | 0 | 0 | 0
Hyperplasia (General disorders) | 1 | 0 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0
Implant site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 2 | 0 | 0 | 1
Multi-organ failure (General disorders) | 3 | 4 | 2 | 6
Non-cardiac chest pain (General disorders) | 45 | 33 | 33 | 46
Oedema (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 3 | 7 | 3
Pain (General disorders) | 1 | 0 | 0 | 1
Pelvic mass (General disorders) | 0 | 0 | 1 | 0
Polyp (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 7 | 9 | 4 | 9
Submandibular mass (General disorders) | 0 | 0 | 0 | 1
Sudden cardiac death (General disorders) | 7 | 6 | 11 | 12
Sudden death (General disorders) | 2 | 1 | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Vestibulitis (General disorders) | 0 | 0 | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1 | 1 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 3
Bile duct stone (Hepatobiliary disorders) | 3 | 4 | 6 | 9
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 8 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary fistula (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Biloma (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 3 | 3 | 3
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 9 | 11 | 12 | 15
Cholecystitis acute (Hepatobiliary disorders) | 10 | 8 | 6 | 8
Cholecystitis chronic (Hepatobiliary disorders) | 10 | 5 | 0 | 2
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 26 | 28 | 48 | 30
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gallbladder cholesterolosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Gallbladder fistula (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 2 | 1 | 1
Hepatic infarction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 3 | 2 | 3 | 5
Jaundice cholestatic (Hepatobiliary disorders) | 4 | 1 | 4 | 1
Jaundice hepatocellular (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Perforation bile duct (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Porcelain gallbladder (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 3 | 1 | 3 | 3
Hypersensitivity (Immune system disorders) | 0 | 1 | 2 | 0
Iodine allergy (Immune system disorders) | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 1 | 0
Abscess (Infections and infestations) | 3 | 2 | 1 | 2
Abscess intestinal (Infections and infestations) | 0 | 1 | 2 | 1
Abscess limb (Infections and infestations) | 2 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 2
Anal abscess (Infections and infestations) | 0 | 1 | 1 | 1
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 4 | 2 | 5 | 9
Appendicitis perforated (Infections and infestations) | 1 | 1 | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 3 | 0 | 0
Arthritis infective (Infections and infestations) | 2 | 2 | 2 | 1
Bacillus infection (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Biliary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Borrelia infection (Infections and infestations) | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 5 | 12 | 8 | 12
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 5 | 6 | 8 | 3
Bursitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Campylobacter intestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 2 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 2 | 1
Catheter sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 14 | 19 | 10 | 13
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis streptococcal (Infections and infestations) | 2 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 1 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 1 | 0 | 1
Chronic sinusitis (Infections and infestations) | 3 | 1 | 3 | 1
Citrobacter infection (Infections and infestations) | 0 | 1 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 0 | 2 | 1
Clostridium difficile sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 2 | 0 | 2
Cystitis escherichia (Infections and infestations) | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 2 | 0 | 1 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 5 | 7 | 7 | 12
Douglas' abscess (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Ear lobe infection (Infections and infestations) | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 5 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 1
Epidemic nephropathy (Infections and infestations) | 1 | 0 | 0 | 0
Epididymal infection (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 6 | 6 | 3 | 5
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 4
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 1
Gallbladder empyema (Infections and infestations) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 1 | 0
Gastric ulcer helicobacter (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 10 | 12 | 6 | 7
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 4 | 4 | 4
Graft infection (Infections and infestations) | 0 | 0 | 2 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 1 | 0 | 1
Hepatitis non-A non-B (Infections and infestations) | 0 | 0 | 0 | 1
Hepatitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 3 | 1 | 2
Herpes zoster infection neurological (Infections and infestations) | 1 | 0 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 1
Incision site infection (Infections and infestations) | 1 | 0 | 0 | 1
Infected bites (Infections and infestations) | 0 | 1 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 3 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 0 | 1 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 2
Injection site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 3 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 2
Lobar pneumonia (Infections and infestations) | 3 | 3 | 2 | 1
Localised infection (Infections and infestations) | 0 | 1 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 5 | 5 | 9 | 10
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 2 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 1
Mediastinitis (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 2
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Miliary pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Morganella infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 2
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Neisseria infection (Infections and infestations) | 0 | 1 | 0 | 0
Neuroborreliosis (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0 | 1 | 0
Peridiverticular abscess (Infections and infestations) | 0 | 0 | 0 | 1
Perihepatic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Peritoneal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0 | 1 | 0
Pleural infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 47 | 33 | 41 | 43
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 2 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 3 | 0
Post procedural infection (Infections and infestations) | 1 | 1 | 5 | 1
Post procedural pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 5 | 2 | 9 | 4
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 3 | 2 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 3 | 1 | 2
Pyelonephritis chronic (Infections and infestations) | 2 | 2 | 0 | 1
Pyothorax (Infections and infestations) | 0 | 0 | 1 | 2
Respiratory tract infection (Infections and infestations) | 2 | 3 | 3 | 2
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1 | 1 | 1
Salpingitis (Infections and infestations) | 0 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 0 | 1 | 1
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 9 | 4 | 9 | 16
Septic embolus (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 5 | 3 | 2 | 0
Shunt infection (Infections and infestations) | 0 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 4 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 2 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Subacute endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Superinfection (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Tularaemia (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 3 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 16 | 14 | 17 | 14
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 8 | 2 | 2 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 2 | 0 | 0
Viral infection (Infections and infestations) | 2 | 1 | 3 | 0
Viral pericarditis (Infections and infestations) | 0 | 1 | 0 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 2 | 1 | 3 | 1
Wound infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 2 | 1
Wound sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Anal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 5 | 5 | 6
Anxiety postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Asbestosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 2
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Cold exposure injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 2 | 5 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 5 | 2 | 3
Corneal scar (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Device breakage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Device malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Drug dose omission (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0
Electric shock (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 3 | 4 | 0 | 2
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 1
Failure of implant (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 46 | 47 | 59 | 36
Fat embolism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3 | 5 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gallbladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 4 | 6 | 8
Hip fracture (Injury, poisoning and procedural complications) | 5 | 5 | 5 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 6 | 2 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 7 | 8 | 3 | 4
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intraocular lens dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 5 | 2 | 4
Joint injury (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 3 | 3 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 4 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 8 | 5 | 2 | 11
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 6 | 2 | 2 | 5
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 5
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 7 | 1 | 0 | 5
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radial nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 3
Renal injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 5 | 4 | 3 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 14 | 7 | 9 | 9
Seroma (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 1
Snake bite (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 1
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 5
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 5 | 2 | 3 | 2
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 1 | 7 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 4 | 4 | 3 | 5
Urinary bladder rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 4 | 4 | 3
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Vertebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 5 | 3 | 4 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Antinuclear antibody increased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood amylase increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0 | 0
Vascular resistance systemic (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 4 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Central obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 12 | 10 | 12 | 15
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 6 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4 | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lipomatosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 3 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 12 | 8 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 9 | 10 | 7
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 14 | 11 | 5
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5 | 4
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 3
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 13 | 12 | 12 | 11
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Joint instability (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 11 | 7 | 4 | 6
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 5 | 4
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 77 | 92 | 92 | 93
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 8 | 7 | 11
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4 | 5
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 7 | 3 | 6 | 8
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Spinal fusion acquired (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 10 | 5 | 6
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 4
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenosquamous cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 16 | 14 | 16
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Benign neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3 | 10
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 3 | 3
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Breast adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 24 | 20 | 14
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1
Chronic lymphocytic leukaemia stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 16 | 13 | 12
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 2
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Endocrine neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 2 | 4
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 7 | 5
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 4 | 3
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intracranial meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 1
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Liposarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 2 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 3 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9 | 16 | 16
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 1
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3 | 3
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Malignant melanoma of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6 | 4 | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 2 | 2
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 7 | 13 | 10
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6 | 4 | 7
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 1 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 2 | 4
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 2 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 3
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Paget's disease of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4 | 2 | 5
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Pharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 | 36 | 34 | 30
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6 | 5 | 5
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 3
Rectal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 3 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 0 | 2
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rosai-Dorfman syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2 | 1 | 5
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 2
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tonsillar neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 3 | 1
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Alcoholic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 3 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 1
Amnestic disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 2 | 0 | 1 | 1
Arachnoid cyst (Nervous system disorders) | 0 | 1 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Basilar artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 2 | 1 | 2
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 4 | 0
Carotid artery stenosis (Nervous system disorders) | 12 | 12 | 16 | 14
Carotid sinus syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 2 | 1
Cataplexy (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebellar atrophy (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebellar haematoma (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 0 | 2 | 0
Cerebral artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 2
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral circulatory failure (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral cyst (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1 | 3 | 3
Cerebral infarction (Nervous system disorders) | 5 | 6 | 4 | 6
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 2 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrospinal fluid rhinorrhoea (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 22 | 34 | 28 | 40
Cerebrovascular disorder (Nervous system disorders) | 1 | 1 | 2 | 2
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 0 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1 | 1 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Coma (Nervous system disorders) | 4 | 1 | 4 | 2
Complex partial seizures (Nervous system disorders) | 1 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 4 | 5 | 5
Coordination abnormal (Nervous system disorders) | 0 | 0 | 2 | 0
Dementia (Nervous system disorders) | 0 | 0 | 5 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 12 | 10 | 13 | 11
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Drop attacks (Nervous system disorders) | 0 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 2 | 2
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 3 | 1
Epilepsy (Nervous system disorders) | 2 | 3 | 3 | 3
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 1 | 1 | 3
Facial paresis (Nervous system disorders) | 1 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 5 | 5 | 4 | 3
Headache (Nervous system disorders) | 5 | 3 | 6 | 4
Hemiparesis (Nervous system disorders) | 2 | 3 | 4 | 2
Hemiplegia (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Horner's syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 2 | 3 | 2 | 2
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 3 | 3
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 2 | 2 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 2 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 2 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 16 | 10 | 13 | 14
Lacunar infarction (Nervous system disorders) | 1 | 2 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2
Leukoaraiosis (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 10 | 9 | 6 | 8
Lumbar radiculopathy (Nervous system disorders) | 0 | 2 | 1 | 2
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1
Morton's neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Multiple system atrophy (Nervous system disorders) | 0 | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1 | 1
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 4
Nerve root compression (Nervous system disorders) | 2 | 0 | 2 | 0
Nerve root lesion (Nervous system disorders) | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 3 | 1 | 5
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 2 | 2 | 1 | 3
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 10 | 10 | 9 | 6
Quadriparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1 | 0 | 1
Radiculitis cervical (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 0 | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 2 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 3 | 3 | 2 | 2
Senile dementia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Spinal claudication (Nervous system disorders) | 3 | 1 | 0 | 2
Spinal cord compression (Nervous system disorders) | 1 | 1 | 2 | 0
Spinal cord ischaemia (Nervous system disorders) | 2 | 0 | 0 | 0
Spinal vascular disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Stupor (Nervous system disorders) | 0 | 0 | 0 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 3 | 3 | 2
Syncope (Nervous system disorders) | 33 | 29 | 26 | 34
Thalamus haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Thoracic outlet syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Tonic convulsion (Nervous system disorders) | 0 | 1 | 1 | 0
Transient global amnesia (Nervous system disorders) | 2 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 26 | 27 | 18 | 24
Tremor (Nervous system disorders) | 0 | 0 | 3 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 2 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 2 | 0 | 2
Vasculitis cerebral (Nervous system disorders) | 0 | 1 | 0 | 0
Vertebral artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Vertebral artery thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 2 | 1 | 2
Wallenberg syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 0 | 2 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 2 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 2 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 4 | 1 | 4
Anxiety disorder (Psychiatric disorders) | 2 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 4 | 3 | 4 | 5
Delirium (Psychiatric disorders) | 0 | 4 | 2 | 1
Delirium tremens (Psychiatric disorders) | 0 | 0 | 1 | 1
Delusion (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 5 | 4 | 5 | 4
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 1
Emotional distress (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 4 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 2 | 2 | 2
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1
Obsessive thoughts (Psychiatric disorders) | 1 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 1 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 2 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 2 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder hypertrophy (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 2 | 1 | 1 | 4
Calculus bladder (Renal and urinary disorders) | 0 | 2 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 4 | 1 | 5 | 3
Calculus urinary (Renal and urinary disorders) | 3 | 1 | 2 | 3
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 2 | 2
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 8 | 7 | 6 | 3
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 4 | 5 | 2
Hydroureter (Renal and urinary disorders) | 0 | 0 | 2 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypotonic urinary bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 1
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 13 | 9 | 11 | 12
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 2 | 1 | 2 | 0
Oliguria (Renal and urinary disorders) | 0 | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 2
Polyuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 1 | 3
Renal atrophy (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 3 | 6 | 5 | 1
Renal cyst (Renal and urinary disorders) | 4 | 1 | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 5 | 11 | 15 | 8
Renal failure acute (Renal and urinary disorders) | 14 | 10 | 11 | 6
Renal failure chronic (Renal and urinary disorders) | 5 | 3 | 1 | 3
Renal impairment (Renal and urinary disorders) | 1 | 1 | 3 | 3
Renal mass (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal pelvis fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 3 | 3 | 1 | 3
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 2
Ureteric perforation (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral caruncle (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 3 | 2 | 2 | 1
Urethral ulcer (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 6 | 4 | 4 | 3
Urinary retention (Renal and urinary disorders) | 6 | 7 | 8 | 6
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1
Vesical fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 3 | 4 | 2
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 19 | 17 | 28 | 27
Breast calcifications (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Cervix inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Colpocele (Reproductive system and breast disorders) | 0 | 2 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 7 | 8 | 1 | 5
Endometrial atrophy (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Mammary duct ectasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 1 | 2 | 0
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Ovarian atrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 5 | 6 | 3 | 4
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 2 | 2
Prostatitis (Reproductive system and breast disorders) | 2 | 1 | 1 | 2
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 6 | 2
Rectocele (Reproductive system and breast disorders) | 2 | 7 | 1 | 4
Testicular infarction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine cervical laceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 3 | 2 | 0 | 3
Uterine prolapse (Reproductive system and breast disorders) | 5 | 5 | 7 | 11
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2 | 1
Vaginal laceration (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 3 | 8 | 2 | 7
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 4
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Anoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 8 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 | 10 | 18 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 3
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 15 | 28 | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 5
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 3
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 9 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 6
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 20 | 17 | 12 | 9
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 7 | 6
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 11 | 8
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5 | 4
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 4
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Activities of daily living impaired (Social circumstances) | 0 | 1 | 0 | 1
Exposure to chemical pollution (Social circumstances) | 0 | 0 | 1 | 0
Victim of crime (Social circumstances) | 0 | 1 | 0 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 5 | 10 | 14 | 13
Aortic aneurysm rupture (Vascular disorders) | 3 | 1 | 1 | 3
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 1 | 0
Aortic intramural haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Aortic rupture (Vascular disorders) | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 4 | 5 | 2 | 3
Arterial disorder (Vascular disorders) | 1 | 0 | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Arterial insufficiency (Vascular disorders) | 1 | 0 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 1 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 5 | 9 | 4 | 3
Arteriosclerosis obliterans (Vascular disorders) | 0 | 0 | 0 | 1
Arteritis (Vascular disorders) | 1 | 0 | 0 | 0
Artery dissection (Vascular disorders) | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 9 | 11 | 11 | 4
Deep vein thrombosis (Vascular disorders) | 12 | 7 | 13 | 13
Diabetic vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 1
Essential hypertension (Vascular disorders) | 1 | 2 | 2 | 4
Exsanguination (Vascular disorders) | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 2 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1 | 1 | 2
Flushing (Vascular disorders) | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 2 | 5 | 0 | 2
Haemodynamic instability (Vascular disorders) | 2 | 1 | 0 | 2
Haemorrhage (Vascular disorders) | 3 | 1 | 0 | 0
Haemorrhagic infarction (Vascular disorders) | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 19 | 15 | 35 | 27
Hypertensive crisis (Vascular disorders) | 12 | 13 | 13 | 10
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 0
Hypoperfusion (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 22 | 19 | 21 | 12
Hypovolaemic shock (Vascular disorders) | 0 | 2 | 4 | 0
Iliac artery embolism (Vascular disorders) | 0 | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 1 | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 2 | 1
Intermittent claudication (Vascular disorders) | 5 | 6 | 11 | 9
Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Leriche syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 5 | 2 | 6 | 4
Peripheral artery aneurysm (Vascular disorders) | 2 | 3 | 2 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 5 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 4 | 5
Poor peripheral circulation (Vascular disorders) | 1 | 1 | 0 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 2 | 1 | 1 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian steal syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1 | 0 | 0
Thromboangiitis obliterans (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 2 | 4
Thrombosis (Vascular disorders) | 1 | 2 | 3 | 1
Varicose vein (Vascular disorders) | 4 | 3 | 5 | 4
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Vasodilatation (Vascular disorders) | 0 | 1 | 0 | 2
Vein pain (Vascular disorders) | 1 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 2 | 0 | 0
Venous occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 2
Venous thrombosis limb (Vascular disorders) | 4 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 160 mg od + Nateglinide 60 mg ac (N=2297) | Valsartan 160 mg od + Placebo Nateglinide (N=2283) | Nateglinide 60 mg ac + Placebo Valsartan (N=2305) | Placebo (N=2316)
Angina pectoris (Cardiac disorders) | 114 | 110 | 125 | 119
Vertigo (Ear and labyrinth disorders) | 106 | 117 | 108 | 100
Cataract (Eye disorders) | 148 | 160 | 146 | 163
Abdominal pain (Gastrointestinal disorders) | 128 | 118 | 134 | 134
Abdominal pain upper (Gastrointestinal disorders) | 142 | 126 | 124 | 126
Constipation (Gastrointestinal disorders) | 108 | 95 | 127 | 135
Diarrhoea (Gastrointestinal disorders) | 305 | 299 | 278 | 277
Dyspepsia (Gastrointestinal disorders) | 142 | 142 | 152 | 147
Nausea (Gastrointestinal disorders) | 197 | 176 | 181 | 193
Fatigue (General disorders) | 234 | 202 | 222 | 228
Non-cardiac chest pain (General disorders) | 120 | 116 | 128 | 126
Oedema peripheral (General disorders) | 228 | 198 | 264 | 284
Bronchitis (Infections and infestations) | 218 | 234 | 249 | 226
Influenza (Infections and infestations) | 301 | 309 | 299 | 315
Nasopharyngitis (Infections and infestations) | 396 | 410 | 408 | 385
Sinusitis (Infections and infestations) | 127 | 122 | 134 | 138
Upper respiratory tract infection (Infections and infestations) | 270 | 274 | 250 | 278
Urinary tract infection (Infections and infestations) | 202 | 190 | 225 | 207
Hypercholesterolaemia (Metabolism and nutrition disorders) | 115 | 122 | 137 | 110
Hypoglycaemia (Metabolism and nutrition disorders) | 455 | 271 | 454 | 251
Arthralgia (Musculoskeletal and connective tissue disorders) | 369 | 377 | 377 | 367
Back pain (Musculoskeletal and connective tissue disorders) | 398 | 358 | 339 | 326
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 158 | 163 | 141 | 151
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 226 | 194 | 224 | 241
Pain in extremity (Musculoskeletal and connective tissue disorders) | 280 | 273 | 275 | 238
Dizziness (Nervous system disorders) | 440 | 379 | 397 | 351
Headache (Nervous system disorders) | 242 | 289 | 306 | 311
Depression (Psychiatric disorders) | 146 | 165 | 169 | 158
Insomnia (Psychiatric disorders) | 117 | 94 | 100 | 115
Cough (Respiratory, thoracic and mediastinal disorders) | 238 | 220 | 234 | 224
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 122 | 124 | 152 | 146
Hypertension (Vascular disorders) | 293 | 302 | 392 | 444
Hypotension (Vascular disorders) | 732 | 717 | 582 | 542

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.